CLINICAL TRIAL: NCT06715111
Title: Effect of Laser Acupuncture on Postnatal Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Gomaa Mostafa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alaa-001234
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Laser Acupuncture; Pelvic Pain; Post Natal
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture (Experimental): included twenty-seven participants whom have postnatal pelvic girdle pain received laser acupuncture over specific acupoints, plus conventional pelvic floor exercises; 30minutes, 3 times/week for consecutive 12 sessions for four weeks
  Interventions: Device: Laser acupuncture; Other: conventional pelvic floor exercise
- conventional pelvic floor exercises (Active Comparator): included twenty-seven participants whom have postnatal pelvic girdle pain received conventional pelvic floor exercises; 30minutes, 3 sessions per week consecutive 12 sessions for four weeks
  Interventions: Other: conventional pelvic floor exercise

INTERVENTIONS:
Device: Laser acupuncture — A study used a laser acupuncture device to deliver treatment to 27 participants in Group A. The device, was designed for high power, non-thermal treatment. The device had a Class IV- high power, non-thermal laser with a wave length of 808-905 and a 650 nm wavelength. It had an ergonomic handpiece, high efficiency aiming beam, and adjustable emission intensity range. The device also included two laser safety goggles, a touchscreen stylus, and a retractable banner. Participants were instructed to relax and accurately detect acupoints before application. The device was adjusted for safety and both participants and researchers wore laser goggles.
  Arms: laser acupuncture
Other: conventional pelvic floor exercise — The study involved participants from groups A and B who underwent conventional pelvic floor exercises for four weeks. The exercises targeted the pubococcygeus, sphincter ani, and urethral musculatures. Participants underwent a warm-up phase with 3-5 minutes of breathing and circulatory exercises, followed by 10 repetitions, 3-5 sets, a 3-5 minute warm-up, 30 minutes of exercises, and a cool-down in five minutes. The exercise program was repeated three times per week for four weeks. Participants were instructed to ensure bladder emptiness, relax, perform contractions and relaxations, squeeze pelvic floor musculatures around the anus and vagina, and maintain contact with the plinth. The cool-down phase involved supervised training for 3-5 minutes of breathing and circulatory exercises.

SUMMARY:
this study was done to evaluate the effect of laser acupuncture on pelvic girdle pain postnatal females' patients.

DETAILED DESCRIPTION:
Postnatal pelvic girdle pain might be addressed as a gynecologic challenge in the 21 century in women of all ages and it frequently occur simultaneously. Various forms of postnatal pelvic girdle pain were aggravated by moderate daily activities. Laser acupuncture is a therapeutic modality focuses on selected acupoints in a safe maneuver

ELIGIBILITY:
Inclusion Criteria:

* Fifty-four women suffering from postnatal pelvic girdle pain, clinically diagnosed by a gynecologist.
* Their ages were ranged from 20-45 years old.
* Their body mass index (BMI) was ranged from 25-29.9 kg/m2.
* They shouldn't have any musculoskeletal or neurological disorders.

Exclusion Criteria:

* Current pregnancy.
* Malignant condition
* History of acute infection
* Neurological problem
* Mental problem to prevent evaluation and cooperation.
* Having uncontrolled metabolic diseases like diabetes and thyroid disease.
* Athletic females.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Fifty-four women suffering from postnatal pelvic girdle pain, clinically diagnosed by a gynecologist.
  * Their ages were ranged from 20-45 years old.
  * Their body mass index was ranged from 25-29.9 kg/m2.
Enrollment: 54 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change of body mass index | At baseline and after 4 weeks
  The study used a method to measure body weight and height of participants in both groups (A & B) to calculate their body mass index, which was calculated by dividing weight in kg by height in m2 for one shot.

SECONDARY OUTCOMES:
Assessment of change of physical activity restrictions | At baseline and after 4 weeks
  The Postnatal Pelvic Girdle Pain Questionnaire was used to assess physical activity restrictions in participants with postnatal pelvic girdle pain before and after treatment. The Postnatal Pelvic Girdle Pain Questionnaire, consisting of 25 items, is a reliable and valid clinical evaluating tool for women with pelvic floor disorders, making it a globally used tool.
Assessment of change of postnatal pelvic girdle pain | At baseline and after 4 weeks
  The Posterior Pelvic Pain Provocation Test was used to assess postnatal pelvic girdle pain in both A&B groups before and after treatment. The test involved a clinician stabilizing the pelvis and applying slight pressure to the femur. A positive Posterior Pelvic Pain Provocation Test was considered if the participant experienced similar pain.
Assessment of change of Salivary Cortisol values | At baseline and after 4 weeks
  Salivary cortisol values were used as an objective biomarker to assess physiologic and psychologic stress associated with postnatal pelvic girdle pain in both groups (A&B) before and after treatment. Saliva was collected before teeth brushing or breaking nocturnal fast, and samples were kept cold and stored at -20°C until laboratory analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Out-patient Clinic of Gynecology department of Mansoura International Hospital, Egypt, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No